CLINICAL TRIAL: NCT04453059
Title: A Phase IIIB, Multicenter Study With Oral Administration of Isovue-300 for Opacification and Delineation of the Gastrointestinal (GI) Tract in Abdominopelvic Computed Tomography (CT)
Brief Title: Study With Oral Isovue in Abdominopelvic CT
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IOP-121
Record Dates: First submitted 2020-06-15; First posted 2020-07-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Patients Requiring Abdominopelvic CT With Oral Administration of Contrast
Keywords: Oral Isovue
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Iopamidol — Previously administered Isovue-300 (300 mgI/mL) PO at a dilution of 2-3% (6-9 mgI/mL)

SUMMARY:
This is a retrospective clinical study with prospectively designed blinded evaluation of CT images in adult and pediatric patients who underwent CT examinations of the abdomen and pelvis and were orally administered a solution of Isovue-300 to opacify the GI tract to distinguish it from adjacent abdominal and pelvic structures. The study will collect already existing data, such as demographic data, adverse events and CT images, for all chronologically enrolled patients who meet the inclusion/exclusion criteria prospectively defined in this protocol

ELIGIBILITY:
Patients will be included in the study if:

* Demographic and safety data are available for analysis
* Complete set of CT images performed after oral administration of Isovue-300 are available for assessment
* Isovue-300 was orally administered during an interval time of 60-20 minutes before the CT scanning.

Patients will be excluded from the study if:

* Oral contrast agent received within 1 week prior to the CT scan
* Undergone any abdominopelvic surgery procedure that resulted in alteration of the bowel transit time prior to the CT exam
* CT exam with oral administration of Isovue was performed because of a known or suspected condition of bowel obstruction
* Patient did not actively drink the contrast solution.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients who have previously undergone CT examination of the abdomen and pelvis with oral administration of Isovue-300 (2-3% concentration) as part of their clinical work-up.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adequate visualization of anatomic delineation of the GI tract | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States